CLINICAL TRIAL: NCT07213128
Title: The Effect of Home-based Inspiratory Muscle Training Compared to Usual Care on Readmission Rate in Patients After a Severe Acute Exacerbation of Chronic Obstructive Pulmonary Disease: a Randomised, Multicentre, Parallel Group Clinical Trial: IN-SPIRED Trial
Brief Title: Effect of IMT in Patients After Acute Exacerbations of COPD
Acronym: IN-SPIRED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Hopitaux Iris Sud (Unknown); Centre Hospitalier Universitaire Saint Pierre (Other); Onze Lieve Vrouw Hospital (Other); AZ Delta (Other); University Hospital, Antwerp (Other); Algemeen Ziekenhuis Maria Middelares (Other); Grand Hôpital de Charleroi (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other); Centre Hospitalier Universitaire de Liege (Other); General Hospital Groeninge (Other); University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Daniel Langer, associate professor Faculty of Movement and Rehabilitation Sciences, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S68174; INV23-1479 (Other: KCE Trials); S68174 (Other: UZ/KU Leuven)
Record Dates: First submitted 2025-09-15; First posted 2025-10-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Diseases; COPD; Symptom Exacerbation
Keywords: Inspiratory muscle training; Respiratory muscle training; acute exacerbation; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Symptom Flare Up

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Training
- Control (No Intervention): Patients will receive usual care, including optimal pharmacological therapy per international guidelines, advise on smoking cessation, vaccination, and physical activity participation and advised to attend physiotherapy or a respiratory rehabilitation program based on accessibility and patient preference.

INTERVENTIONS:
Other: Training — home-based inspiratory muscle training (IMT) will be delivered using a portable IMT device connected via Bluetooth to a smartphone application that provides real-time feedback, adherence monitoring, and telemonitoring by the study team. Patients will train for 365 days following hospital discharge due to an acute exacerbation of COPD:
  * Intensive phase (Day 0-90): 2 daily sessions, each consisting of 30 breaths against an inspiratory load set by thetelemonitor, with regular online supervised IMT sessions, 7 sessions in total
  * Maintenance phase (Day 91-180): One daily session of 30 breaths, with sporadic online supervised IMT sessions, 2 sessions in total.
  * Follow-up phase (Day 181-365): Participants may continue IMT unsupervised. Supervision includes both in-person sessions at hospital visits and online sessions with telemonitors.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test whether home-based inspiratory muscle training can reduce hospital readmissions and death in patients recovering from a severe acute exacerbation of chronic obstructive pulmonary disease (AECOPD).

The main questions this study aims to answer are:

Does adding home-based inspiratory muscle training to usual care lower the risk of all-cause hospital readmission or death within 180 days after discharge? Does inspiratory muscle training improve respiratory muscle strength, symptoms of dyspnea, quality of life, and functional capacity compared to usual care?

Researchers will compare patients randomized to:

Intervention group: Home-based inspiratory muscle training plus usual care Control group: Usual care only

to see if inspiratory muscle training leads to fewer readmissions and deaths, and better patient-reported and physiological outcomes.

Participants will:

Be hospitalized for ≥3 days due to AECOPD, age ≥35 years, able to consent, and own a compatible smartphone.

In the intervention group, receives usual care and additionally inspiratory muscle training:

Inspiratory muscle training twice daily for 90 days, then once daily up to day 180, with remote telemonitoring via a smartphone app and online supervised sessions.

The control group will continue with usual care (pharmacological treatment, smoking cessation advice, vaccinations, and referral to pulmonary rehabilitation if available).

Follow-up assessments will include hospital readmissions, survival, and quality of life questionnaires up to 12 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the hospital ≥3 days for AECOPD
* Read and speak French, Dutch or English
* Age ≥ 35 years
* Able to provide informed consent
* Possessing a smartphone, compatible with the tele-monitoring app and able to perform video meetings.

Exclusion Criteria:

* Patients already performing IMT at time of inclusion
* Patients with estimated <90 days life expectancy
* Non-COPD pulmonary disease as primary diagnosis
* Active malignancy
* Inability to perform IMT or response to questionnaires (e.g., neurological/cognitive impairment)
* Acute instable cardiac arrythmia or ischemia
* Acute pneumothorax
* Planned lung volume reduction procedure <180days
* Waitlisted for lung transplantation
* Patients admitted to an in-hospital rehabilitation ward
* Patients included in other interventional trial related to COPD that would interfere with our trial outcomes.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Composite outcome (all-cause hospital readmission or mortality) | within 180 days after hospital discharge

SECONDARY OUTCOMES:
Composite outcome (all-cause hospital readmission or mortality) | within 90 days after hospital discharge
  Occurrence
Time-to-composite outcome (all-cause hospital readmission or mortality) | within 180 days after hospital discharge
  Time-to-event
Hospital re-admission | Day 28, 90 and 180 after hospital discharge
  1. Occurrence
  2. Reason
All-cause mortality | Day 28, 90 and 180 after hospital discharge
  1. Occurrence
  2. Reason
Primary care and specialty consultationsc | Day 90 and 180 after hospital discharge
  Number of days post-discharge
Re-exacerbation | Day 90 and 180 after hospital discharge
  1. Occurrence
  2. Number of occurrences/patient post-discharge
Change in Forced Expiratory Volume in 1 Second (FEV₁), liters | Day 90 and 180 after hospital discharge
  - Mean change in FEV₁ (liters) from baseline, measured by spirometry, according to ATS/ERS guidelines.
Change in Forced Expiratory Volume in 1 Second (FEV₁), %pred | Day 90 and 180 after hospital discharge
  - Mean change in FEV₁ (% predicted) from baseline, measured by spirometry.
Change in Forced Vital Capacity (FVC), liters | Day 90 and Day 180 after hospital discharge
  - Mean change in FVC (liters) from baseline, measured by spirometry.
Change in Forced Vital Capacity (FVC), %predicted | Day 90 and Day 180 after hospital discharge
  - Mean change in FVC (% predicted) from baseline, measured by spirometry.
Change in FEV₁/FVC Ratio (%) | Day 90 and Day 180 after hospital discharge
  Mean change in the ratio of FEV₁ to FVC (percentage) from baseline, measured by spirometry.
Change in Functional Residual Capacity (FRC), liters | Day 180 after hospital discharge
  - Mean change in FRC (liters) from baseline, measured by body plethysmography.
Change in Functional Residual Capacity (FRC), %predicted | Day 180 after hospital discharge
  - Mean change in FRC (% predicted) from baseline, measured by body plethysmography.
Change in Residual Volume (RV), liters | Day 180 after hospital discharge
  - Mean change in RV (liters) from baseline, measured by body plethysmography.
Change in Residual Volume (RV), % predicted | Day 180 after hospital discharge
  - Mean change in RV (% predicted) from baseline, measured by body plethysmography.
Change in Total Lung Capacity (TLC), liters | Day 180 after hospital discharge
  - Mean change in TLC (liters) from baseline, measured by body plethysmography.
Change in Total Lung Capacity (TLC), %predicted | Day 180 after hospital discharge
  - Mean change in TLC (% predicted) from baseline, measured by body plethysmography.
Maximal inspiratory pressure (PImax) | Day 90 and 180 after hospital discharge
  Change from baseline
Baseline/Transition Dyspnea Index (BDI/TDI) | Day 28, 90, 180 after hospital discharge
  Change from baseline
EQ-5D-5L questionnaire | Day 28, 90, 180 after hospital discharge
  Change from baseline
COPD Assessment test (CAT) | Day 28, 90, 180 after hospital discharge
  Change from baseline
Adverse events | Day 90, 180 after hospital discharge
  1. Occurrence
  2. Number of occurrences/patient post-discharge
Serious adverse events | Day 90 and 180 after hospital discharge
  1. Occurrence
  2. Number of occurrences/patient post-discharge

OTHER OUTCOMES:
Intensive care unit admission | Day 90, 180, 365 after hospital discharge
  Number of days post-discharge
Lung function: Diffusion capacity | Day 180 after hospital discharge
  Mean of 2 acceptable assessments
1 minute sit-to-stand test, Repetitions from Baseline | Day 180 after hospital discharge
  Mean change in the number of repetitions completed in the 1-minute sit-to-stand test compared with baseline.
Number of Participants Achieving the Minimal Important Difference (MID) in the 1-Minute Sit-to-Stand Test | Day 180 after hospital discharge
  Number of participants who improved their 1-minute sit-to-stand repetitions by more than the minimal important difference (MID)
Hospital Anxiety & Depression Scale (HADS) | Day 90 and 180 after hospital discharge
  Change from baseline
EQ-5D-5L | Day 365 after hospital discharge
  Change from baseline
COPD Assessment test (CAT) | Day 365 after hospital discharge
  Change from baseline
Baseline/Transition Dyspnea Index (BDI/TDI) | Day 365 after hospital discharge
  Change from baseline
Hospital re-admission | Day 365 after hospital discharge
  Time to event
All-cause mortality | Day 365 after hospital discharge
  1. Time to event
  2. Reason
Rate of AECOPD treated with systemic corticosteroids | Day 90, 180, 365 after hospital discharge
  1. Occurrence
  2. Time to event
Rate of AECOPD treated with antibiotics | Day 90, 180, 365 after hospital discharge
  1. Occurrence
  2. Time to event

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Langer, PhD, Principal Investigator — KU Leuven
Locations (12):
- Belgium (12):
  - AZORG, Aalst
  - Campus Joseph Bracops, Hôpitaux Iris Sud, Anderlecht
  - Centre Hospitalier Universitaire Saint-Pierre, Brussels
  - Grand Hopial de Charleroi, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge, Kortrijk
  - University Hospitals Leuven, Leuven
  - Centre hospitalier universitaire de Liège, Liège
  - AZ Delta, Roeselare
  - Centre Hospitalier Universitaire UCL Namur, Yvoir

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share individual participant data (IPD). De-identified participant-level data will not be made publicly available. However, summary results of the trial will be published in peer-reviewed journals and presented at scientific meetings. Researchers interested in secondary analyses may contact the sponsor (UZ Leuven) to discuss possibilities for collaborative projects, subject to approval by the Trial Steering Committee and compliance with applicable regulations and GDPR.